CLINICAL TRIAL: NCT02505828
Title: ARTEMIS Synovial Markers in Arthritis Childhood
Acronym: ARTEMIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 93612; 2014-A01561-46 (Registry Identifier: ID RCB)
Record Dates: First submitted 2015-06-22; First posted 2015-07-22 (Estimated); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Septic Arthritis; Juvenile Idiopathic Arthritis
Keywords: Arthritis; septic; Juvenile idiopathic arthritis; diagnosis; proteomic; cytokine; monocytes
MeSH Terms: conditions — Arthritis, Infectious; Arthritis, Juvenile; Arthritis; Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Septic arthritis (Other): with bacteriological identification
  Interventions: Procedure: Articular punction, salivary samples, blood sample
- Juvenile idiopathic arthritis (Other): beyond the ILAR (International League of Associations for Rheumatology) definition
  Interventions: Procedure: Articular punction, salivary samples, blood sample

INTERVENTIONS:
Procedure: Articular punction, salivary samples, blood sample
  Other Names: Proteomic analysis; Cytokine dosage; Monocyte

SUMMARY:
The aim of this study is to find markers that could differentiate infectious and inflammatory arthritis. The investigators want to find markers by differential analysis by compare synovial fluids of septic and inflammatory arthritis. The investigators will use for this analysis, proteomics, cytokine dosage and monocyte typing by flow cytometry analysis. The investigators will use one marker or a score with biological and clinical data to discriminate arthritis of infectious and inflammatory etiology.

ELIGIBILITY:
Inclusion Criteria:

* Septic arthritis with bacteriological identification
* Juvenile idiopathic arthritis beyond the ILAR definition
* Having acute arthritis requiring an articular draining
* Child benefiting from a national insurance scheme
* Collection of the consent of the parents or the legal representative

Exclusion Criteria:

* Contraindication in an articular draining: platelet 50 000 / mm3, Rate of prothrombins lower than 70 %, activated partial thromboplastin times (APTT)> 1,5
* Treatment by biotherapy, corticoids or other immuno suppressor in the month preceding the articular draining.
* Treatment by antibiotic begun more than 24 hours before the draining.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2015-04; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Qualitative analysis of new biological markers (proteic, cytokine or cellular) that discriminate inflammatory and infectious arthritis. | 1 day
  Identify blood sampling biomarkers of Arthritis childhood

CONTACTS AND LOCATIONS:
Overall Officials: Eric EJ JEZIORSKI, MD, PhD, Principal Investigator — Montpellier University Hospital
Locations (1):
- Hôpital Arnaud de Villeneuve, Montpellier, France

REFERENCES:
- [Result] Nziza N, Jeziorski E, Delpont M, Cren M, Chevassus H, Carbasse A, Mahe P, Abassi H, Joly-Monrigal P, Schordan E, Mange A, Jorgensen C, Apparailly F, Duroux-Richard I. Synovial-Fluid miRNA Signature for Diagnosis of Juvenile Idiopathic Arthritis. Cells. 2019 Nov 26;8(12):1521. doi: 10.3390/cells8121521. PMID 31779271
- [Result] Cren M, Nziza N, Carbasse A, Mahe P, Dufourcq-Lopez E, Delpont M, Chevassus H, Khalil M, Mura T, Duroux-Richard I, Apparailly F, Jeziorski E, Louis-Plence P. Differential Accumulation and Activation of Monocyte and Dendritic Cell Subsets in Inflamed Synovial Fluid Discriminates Between Juvenile Idiopathic Arthritis and Septic Arthritis. Front Immunol. 2020 Jul 31;11:1716. doi: 10.3389/fimmu.2020.01716. eCollection 2020. PMID 32849606